CLINICAL TRIAL: NCT02979964
Title: Pragmatic Factorial Cluster Trial of Framing and Comparators for Audit and Feedback Aiming to Address High Risk Prescribing in Nursing Homes in Ontario
Brief Title: Pragmatic Factorial Cluster Trial of Framing and Comparators for Audit and Feedback
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Women's College Hospital (Other)
Collaborators: Health Quality Ontario (Other)
Responsible Party: Principal Investigator, Noah Ivers, M.D., PhD, CCFP, Women's College Hospital
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2016-0122-E
Record Dates: First submitted 2016-11-29; First posted 2016-12-02 (Estimated); Last update posted 2018-10-05 (Actual); Status verified 2018-10

CONDITIONS: High-risk Prescribing in Nursing Homes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1, Positive Framing (Experimental): All metrics in the audit and feedback practice reports presented with 'positive' framing, where the proportion of patients safe from risk (i.e., appropriate/desirable prescribing behaviours) is described.
  Interventions: Behavioral: Audit and Feedback
- Arm 2, Negative Framing (Experimental): All metrics in the audit and feedback practice reports presented with 'negative' framing, where the proportion of patients at risk (i.e., due to inappropriate/undesirable prescribing behaviours) is described.
  Interventions: Behavioral: Audit and Feedback
- Arm 3, Top Quartile Comparator (Experimental): All metrics in the audit and feedback practice reports presented and the physician-recipient's performance is compared against the 75th percentile for performance by physicians working in nursing homes in the province for each metric.
  Interventions: Behavioral: Audit and Feedback
- Arm 4, Average Comparator (Experimental): All metrics in the audit and feedback practice reports presented and the physician-recipient's performance is compared against the average performance by physicians working in nursing homes in the province for each metric.
  Interventions: Behavioral: Audit and Feedback

INTERVENTIONS:
Behavioral: Audit and Feedback

SUMMARY:
Health Quality Ontario (HQO) is the provincial advisor on quality in health care. HQO currently conducts audit and feedback as a key quality improvement strategy. For example, it offers physicians working in long-term care homes with access to practice reports detailing rates of high-risk prescribing in comparison with others in Ontario and suggested change ideas. Research shows that providing this kind of feedback can lead to improvements in care. However, the size of these improvements depends how the feedback is presented. For instance, prior research suggests that how the results are 'framed' and what sort of benchmark the recipient is compared to may each affect how the physician will respond. This factorial trial tests each of these aspects of feedback design in the context of practice reports that nursing home physicians have already signed up to receive quarterly.

ELIGIBILITY:
Inclusion Criteria:

* a physician licensed by the College of Physicians and Surgeons of Ontario (CPSO);
* practice in at least one LTC facility in Ontario;.
* have voluntarily signed up to receive an HQO practice report

Exclusion Criteria:

* n/a

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 285 (Actual)
Dates: Start 2016-12-06 (Actual); Primary Completion 2017-10-06 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
CNS-active medication prescribing | 6 months
  monthly number of CNS-active medications per resident (antipsychotics, opioids, benzodiazepines or antidepressants (including TCAs and trazodone))

SECONDARY OUTCOMES:
Benzodiazepine (or z-drug) prescribing | 6 months
  days supplied (continuous)
Benzodiazepine (or z-drug) rates | 6 months
  monthly proportion
Antipsychotic rates | 6 months
  monthly proportion
Antipsychotic prescribing | 6 months
  days supplied (continuous)
Mean Antipsychotic dose | 6 months
  Dose equivalent of antipsychotic dispensed (continuous)
Mean Benzodiazepine dose | 6 months
  Dose equivalent of benzodiazepine dispensed (continuous)
3+ CNS-active medications | 6 months
  monthly proportion supplied three or more meds from the following classes: antipsychotics, opioids, benzodiazepines, or antidepressants (including TCAs and trazodone).
Anti-depressant prescribing | 6 months
  days supplied (continuous) - balance measure
Anti-acid prescribing | 6 months
  days supplied (continuous) - tracer outcome
Statin prescribing | 6 months
  days supplied (continuous) - tracer outcome

CONTACTS AND LOCATIONS:
Overall Officials: Noah M Ivers, MD PhD CCFP, Principal Investigator — Women's College Hospital - University of Toronto
Locations (1):
- Women's College Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Analyses of outcomes use routine administrative database holdings.

REFERENCES:
- [Background] Ivers NM, Sales A, Colquhoun H, Michie S, Foy R, Francis JJ, Grimshaw JM. No more 'business as usual' with audit and feedback interventions: towards an agenda for a reinvigorated intervention. Implement Sci. 2014 Jan 17;9:14. doi: 10.1186/1748-5908-9-14. PMID 24438584
- [Background] Ivers N, Jamtvedt G, Flottorp S, Young JM, Odgaard-Jensen J, French SD, O'Brien MA, Johansen M, Grimshaw J, Oxman AD. Audit and feedback: effects on professional practice and healthcare outcomes. Cochrane Database Syst Rev. 2012 Jun 13;2012(6):CD000259. doi: 10.1002/14651858.CD000259.pub3. PMID 22696318
- [Background] Kiefe CI, Allison JJ, Williams OD, Person SD, Weaver MT, Weissman NW. Improving quality improvement using achievable benchmarks for physician feedback: a randomized controlled trial. JAMA. 2001 Jun 13;285(22):2871-9. doi: 10.1001/jama.285.22.2871. PMID 11401608
- [Background] Akl EA, Oxman AD, Herrin J, Vist GE, Terrenato I, Sperati F, Costiniuk C, Blank D, Schunemann H. Framing of health information messages. Cochrane Database Syst Rev. 2011 Dec 7;(12):CD006777. doi: 10.1002/14651858.CD006777.pub2. PMID 22161408
- [Background] Kluger AN, Van Dijk D. Feedback, the various tasks of the doctor, and the feedforward alternative. Med Educ. 2010 Dec;44(12):1166-74. doi: 10.1111/j.1365-2923.2010.03849.x. PMID 21091758
- [Background] Hibbard JH, Peters E, Slovic P, Finucane ML, Tusler M. Making health care quality reports easier to use. Jt Comm J Qual Improv. 2001 Nov;27(11):591-604. doi: 10.1016/s1070-3241(01)27051-5. PMID 11708039
- [Background] Gould NJ, Lorencatto F, Stanworth SJ, Michie S, Prior ME, Glidewell L, Grimshaw JM, Francis JJ. Application of theory to enhance audit and feedback interventions to increase the uptake of evidence-based transfusion practice: an intervention development protocol. Implement Sci. 2014 Jul 29;9:92. doi: 10.1186/s13012-014-0092-1. PMID 25070404
- [Background] Weissman NW, Allison JJ, Kiefe CI, Farmer RM, Weaver MT, Williams OD, Child IG, Pemberton JH, Brown KC, Baker CS. Achievable benchmarks of care: the ABCs of benchmarking. J Eval Clin Pract. 1999 Aug;5(3):269-81. doi: 10.1046/j.1365-2753.1999.00203.x. PMID 10461579
- [Background] Li AC, Kannry JL, Kushniruk A, Chrimes D, McGinn TG, Edonyabo D, Mann DM. Integrating usability testing and think-aloud protocol analysis with "near-live" clinical simulations in evaluating clinical decision support. Int J Med Inform. 2012 Nov;81(11):761-72. doi: 10.1016/j.ijmedinf.2012.02.009. Epub 2012 Mar 27. PMID 22456088
- [Background] Cane J, O'Connor D, Michie S. Validation of the theoretical domains framework for use in behaviour change and implementation research. Implement Sci. 2012 Apr 24;7:37. doi: 10.1186/1748-5908-7-37. PMID 22530986
- [Derived] McCleary N, Desveaux L, Presseau J, Reis C, Witteman HO, Taljaard M, Linklater S, Thavorn K, Dobell G, Mulhall CL, Lam JMC, Grimshaw JM, Ivers NM. Engagement is a necessary condition to test audit and feedback design features: results of a pragmatic, factorial, cluster-randomized trial with an embedded process evaluation. Implement Sci. 2023 May 10;18(1):13. doi: 10.1186/s13012-023-01271-6. PMID 37165413
- [Derived] Ivers NM, Desveaux L, Presseau J, Reis C, Witteman HO, Taljaard MK, McCleary N, Thavorn K, Grimshaw JM. Testing feedback message framing and comparators to address prescribing of high-risk medications in nursing homes: protocol for a pragmatic, factorial, cluster-randomized trial. Implement Sci. 2017 Jul 14;12(1):86. doi: 10.1186/s13012-017-0615-7. PMID 28705208
- See also: Health Quality Ontario Long-Term Care Practice Report — http://www.hqontario.ca/Quality-Improvement/Practice-Reports/Long-Term-Care